CLINICAL TRIAL: NCT06672640
Title: Effects of Remote Exercise on Physical Function in Pre-Frail Older Adults: A Randomized Controlled Trial
Brief Title: Effects of Remote Exercise on Physical Function in Pre-Frail Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungdong University (Other)
Responsible Party: Principal Investigator, Kyeongjin Lee, professor, Kyungdong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-05-014
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Frail Elderly
Keywords: Telerehabilitation; Postural balance; Gait; Frail Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluators were blinded to the intervention details of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- remote exercise group (Experimental): Participants in the remote exercise group will engage in exercise sessions conducted twice weekly for eight weeks using video conferencing software. The intervention includes balance, strength, and gait training, supervised by a licensed physical therapist. Sessions are performed at participants' homes with assistance from caregivers to ensure safety and compliance.
  Interventions: Behavioral: Remote Exercise Program
- in-person exercise group (Experimental): Participants in the in-person exercise group will attend supervised exercise sessions at a senior welfare center twice weekly for eight weeks. The sessions, conducted by a licensed physical therapist, focus on improving balance, lower limb strength, and gait stability. The intervention is identical to the remote exercise group, except the mode of delivery is in person at the welfare center.
  Interventions: Behavioral: In-Person Exercise Program
- control group (Other): Participants in the control group will receive an informational booklet on exercise and attend a single educational session about physical activity. They will be encouraged to maintain their usual activities, and their physical activity levels will be self-reported and periodically monitored by the research team.
  Interventions: Other: Physical Activity Education

INTERVENTIONS:
Behavioral: Remote Exercise Program — Participants in this group will engage in an eight-week exercise program conducted via video conferencing software. The sessions, which focus on balance, lower limb strength, and gait function, will be held twice weekly for 50 minutes each. Licensed physical therapists will supervise the sessions, and participants will exercise at home, with assistance from caregivers if necessary. The program aims to evaluate the effectiveness of remote exercise interventions in improving physical function and reducing the risk of falls in pre-frail older adults.
  Arms: remote exercise group
Behavioral: In-Person Exercise Program — Participants in this group will take part in an eight-week in-person exercise program at a senior welfare center. The sessions will be held twice weekly for 50 minutes and will be led by a licensed physical therapist. The exercise program, which includes balance, lower limb strength, and gait training, is identical to that of the remote exercise group, with the primary difference being the mode of delivery (in-person at the welfare center). This group aims to assess the effectiveness of direct supervision in a controlled environment.
  Arms: in-person exercise group
Other: Physical Activity Education — Participants in this group will receive educational materials about physical activity, including a booklet and one educational session. They will not participate in any structured exercise program but will be encouraged to maintain their usual activities. The control group serves as a baseline to compare the outcomes of exercise interventions against no structured exercise, focusing on evaluating usual care versus targeted exercise programs.
  Arms: control group

SUMMARY:
This study aims to compare the effects of remote versus in-person exercise interventions on physical function, balance, gait stability, and fall efficacy in pre-frail older adults aged 65 years and above. Participants are randomly assigned to either a remote exercise group, an in-person exercise group, or a control group. The exercise intervention includes balance, strength, and gait training conducted twice weekly for eight weeks. The control group receives educational materials on physical activity. The primary outcome measures include assessments of balance, lower limb strength, gait ability, and fall efficacy. This study seeks to determine if remote exercise is as effective as in-person exercise in enhancing physical function in pre-frail older adults, potentially providing a feasible alternative to traditional in-person programs and addressing barriers such as limited mobility and access to exercise facilities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Classified as pre-frail based on Fried's frailty criteria (meeting at least two out of five specified indicators)
* Experienced a fall in the preceding six months or have impaired gait and balance (TUG ≥ 13.5 seconds, BBS ≤ 45)
* Mini-Mental State Examination (MMSE) score of 24 or higher
* Demonstrate the physical capacity to engage in the remote exercise (e.g., ability to stand from a seated position and walk short distances)

Exclusion Criteria:

* Neurological or musculoskeletal conditions that impede physical activity
* Recent history of severe cardiovascular disease (within the past three months)
* Inability to commit to continuous participation throughout the study period
* Any other medical condition that might interfere with the intervention or pose a risk to the participant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Balance ability | Baseline and post-intervention at 8 weeks
  Balance performance will be assessed using the Timed Up and Go (TUG) test and Berg Balance Scale (BBS). The TUG measures the time taken for a participant to stand up from a chair, walk three meters, turn around, walk back, and sit down. The BBS is a comprehensive assessment of balance ability during various tasks.
Lower Limb Strength | Baseline and post-intervention at 8 weeks
  Lower limb strength will be evaluated using the Five Times Sit-to-Stand Test (FTSTS) and the 30-Second Chair Stand Test (30SCS). The FTSTS measures the time it takes for participants to rise from a chair five times, and the 30SCS measures the number of times participants can rise from a chair in 30 seconds.
Gait Ability | Baseline and post-intervention at 8 weeks
  Gait ability will be assessed using the Dynamic Gait Index (DGI) and the 10-Meter Walk Test (10MWT). The DGI assesses participants' ability to modify balance while walking in response to external demands, and the 10MWT measures the time taken to walk 10 meters at a comfortable speed.
Fall Efficacy | Baseline and post-intervention at 8 weeks
  Fall efficacy will be measured using the Modified Falls Efficacy Scale (MFES). This scale evaluates participants' confidence in performing daily activities without falling, providing an indication of fall-related self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Kyungdong University, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No